CLINICAL TRIAL: NCT04559347
Title: Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivicaine) Versus Continuous Erector Spinae Plane Block Catheter in Patients Undergoing Video Assisted Thoracoscopic (VAT) Surgery; Single Center, Non Inferiority, Open Label, Randomized Trial
Brief Title: Local Anesthetic as Single Shot Versus Catheter in Patients Undergoing Video Assisted Thoracoscopic Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Poovendran Saththasivam (Other)
Responsible Party: Sponsor-Investigator, Poovendran Saththasivam, Sponsor-Investigator, The Guthrie Clinic
Organization: The Guthrie Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-48
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Surgery
Keywords: Thoracic surgery
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Compare Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine (a long acting local anesthetic) to Ropivacaine (0.5% followed by 0.2% infusion using a catheter) in patients undergoing video assisted thoracoscopic (VAT) surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine (Experimental): Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine for erector spinae block as local anesthetic
  Interventions: Drug: Liposomal Bupivacaine (EXPAREL®)/Bupivacaine
- Continuous catheter infusion ropivacaine (Active Comparator): Ropivacaine (0.5% bolus followed by 0.2% infusion) using a continuous catheter for erector spinae plane block as local anesthetic
  Interventions: Drug: Ropivacaine (0.5% bolus followed by 0.2% infusion)

INTERVENTIONS:
Drug: Liposomal Bupivacaine (EXPAREL®)/Bupivacaine — Single shot for erector spinae block
  Other Names: EXPAREL®/Bupivacaine
  Arms: Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine
Drug: Ropivacaine (0.5% bolus followed by 0.2% infusion) — Continuous catheter infusion for erector spinae plane block
  Other Names: Ropivacaine
  Arms: Continuous catheter infusion ropivacaine

SUMMARY:
The purpose of this research is to compare a single shot long acting local anesthetic to catheter infusion of local anesthetic in patients undergoing video assisted thoracoscopic (VAT) surgery.

DETAILED DESCRIPTION:
The purpose of this research is to compare Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine (a long acting local anesthetic) to Ropivacaine (0.5% bolus followed by 0.2% infusion of local anesthetic using a catheter) in patients undergoing video assisted thoracoscopic (VAT) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are age > 18, undergoing video thoracoscopic surgery and following Guthrie Robert Packer Hospital's Enhanced Recovery After Surgery (ERAS) protocol for Thoracic Surgery.

Exclusion Criteria:

* weight < 50 kg, pregnant subjects,
* left ventricular ejection fraction < 30%,
* history of drug or narcotic abuse,
* history of allergic to amide local anesthetic,
* presence of contraindication for erector spinae plane block (local skin infection, sepsis, severe coagulopathy)
* unable to provide consent,
* unable to use pain rating scales as demonstrated by verbal feedback
* preoperative chronic pain on narcotics,
* history of renal insufficiency ( Creatinine > 1.5 mg/dl),
* preoperative mild liver impairment ( i.e. AST/ALT above 1.5 times the upper normal limit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Poovendran Saththasivam, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Started | 23 | 22
Completed | 17 | 19
Not Completed | 6 | 3
Not completed — Death | 1 | 0
Not completed — Thoracotomy conversion | 1 | 1
Not completed — Provider unavailable | 2 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Due to per protocol analysis for the noninferiority study, the number analyzed differs from the number randomized.
  For the group Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine: 23 subjects were randomized but only 19 subjects received the assignment and only 17 subjects met compliance with protocol to include in final analysis.
  For the Continuous Catheter Infusion Ropivacaine group: 22 subjects were randomized but only 19 met compliance with the protocol to include in final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to per protocol analysis for the noninferiority study, the number analyzed differs from the number randomized. For the Exparel group: 23 subjects were randomized but only 17 subjects complied with protocol to include in final analysis.For the continuous catheter bupivacaine group: 22 subjects were randomized but only 19 complied with the protocol to include in final analysis.
  For the safety analysis of adverse events, all 45 subjectswere included in the analysis.
  years | 65.53 (9.45) | 65.21 (12.91) | 65.36 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 7 | 11 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36
Tobacco History [Count of Participants; unit: Participants]
  Quit more than 12 months ago | 7 | 12 | 19
  Never | 7 | 5 | 12
  Current | 3 | 2 | 5
Chronic liver disease (CLD) history [Count of Participants; unit: Participants] | 0 | 0 | 0
Chronic obstructive pulmonary disease (COPD) History [Count of Participants; unit: Participants] | 0 | 0 | 0
Diabetes History [Count of Participants; unit: Participants] | 2 | 1 | 3
American Society of Anesthesiologists (ASA) Physical Status [Count of Participants; unit: Participants] — The American Society of Anesthesiology (ASA) Physical Status is used to assess a patient's pre-anesthesia medical condition and helps predict how patients will do during a surgical procedure. A lower ASA score predicts (but does not guarantee) better outcomes during a surgical procedure.
  * ASA 1 - a normal healthy patient;
  * ASA 2 - a patient with mild systemic disease;
  * ASA 3 - a patient with severe systemic disease;
  * ASA 4 - a patient with severe systemic disease that is a constant threat to life.
  Participants
    2 | 3 | 3 | 6
    3 | 13 | 16 | 29
    4 | 1 | 0 | 1
Primary Procedure [Count of Participants; unit: Participants]
  Video-assisted thoracoscopic surgery (VATS) with Lobectomy | 12 | 10 | 22
  Video-assisted thoracoscopic surgery (VATS) with Wedge Biopsy | 3 | 7 | 10
  Video-assisted thoracoscopic surgery (VATS) | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rated Pain Scale at Rest 0-4 Hours Post-operative
Description: Patient reported pain scale (0-10) with zero (0) meaning "no pain" and ten (10) meaning "the worst pain imaginable
Time Frame: 0-4 hours post operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 17
score on a scale | 4.824 (2.531) | 5.176 (2.744)

2. Primary Outcome: Numeric Rated Pain Scale at Rest 4-8 Hours Post-operative
Description: Patient reported pain scale (0-10) with zero (0) meaning "no pain" and ten (10) meaning "the worst pain imaginable
Time Frame: 4-8 hours post operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 15 | 15
score on a scale | 3.867 (2.774) | 3.133 (2.386)

3. Primary Outcome: Numeric Rated Pain Scale at Rest 8-12 Hours Post-operative
Description: Patient reported pain scale (0-10) with zero (0) meaning "no pain" and ten (10) meaning "the worst pain imaginable
Time Frame: 8-12 hours post operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 13 | 15
score on a scale | 2.923 (2.253) | 3.4 (2.384)

4. Primary Outcome: Numeric Rated Pain Scale at Rest 12-24 Hours Post-operative
Description: Patient reported pain scale (0-10) with zero (0) meaning "no pain" and ten (10) meaning "the worst pain imaginable
Time Frame: 12-24 hours post operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 14 | 16
score on a scale | 3.714 (2.367) | 5.312 (3.114)

5. Primary Outcome: Numeric Rated Pain Scale at Rest 24-48 Hours Post-operative
Description: Patient reported pain scale (0-10) with zero (0) meaning "no pain" and ten (10) meaning "the worst pain imaginable
Time Frame: 2 days post operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 16 | 16
score on a scale | 4.188 (2.482) | 4.125 (2.187)

6. Primary Outcome: Numeric Rated Pain Scale 48-72 Hours Post-operative
Description: Patient reported pain scale (0-10) with zero (0) meaning "no pain" and ten (10) meaning "the worst pain imaginable
Time Frame: 3 days post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 9 | 6
score on a scale | 3.333 (2.179) | 4.833 (2.639)

7. Primary Outcome: Numeric Rated Pain Scale With Cough 0-4 Hours Post-operative
Description: Patient reported pain with cough on a scale (0-10) with zero (0) meaning "no pain" and ten (10) meaning "the worst pain imaginable
Time Frame: 0-4 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 17
score on a scale | 6.765 (2.306) | 7 (2.784)

8. Primary Outcome: Numeric Rated Pain Scale With Cough 4-8 Hours Post-operative
Description: as for outcome 7
Time Frame: 4-8 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 15 | 14
score on a scale | 7 (2.171) | 5.357 (2.872)

9. Primary Outcome: Numeric Rated Pain Scale With Cough 8-12 Hours Post-operative
Description: as for outcome 7
Time Frame: 8-12 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 13 | 15
score on a scale | 6.615 (2.534) | 5.867 (2.85)

10. Primary Outcome: Numeric Rated Pain Scale With Cough 12-24 Hours Post-operative
Description: as for outcome 7
Time Frame: 12-24 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 15 | 16
score on a scale | 7.467 (2.2) | 7.062 (2.435)

11. Primary Outcome: Numeric Rated Pain Scale With Cough 24-48 Hours Post-operative
Description: as for outcome 7
Time Frame: 24-48 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 16 | 16
score on a scale | 6.875 (2.391) | 7.5 (2.309)

12. Primary Outcome: Numeric Rated Pain Scale With Cough 48-72 Hours Post-operative
Description: as for outcome 7
Time Frame: 48-72 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 9 | 6
score on a scale | 6.889 (2.667) | 6.833 (2.563)

13. Secondary Outcome: Opioid Consumption in Morphine Equivalent Dose 0-4 Hours Post-operative
Description: Post-operative opioid consumption in morphine equivalent dose (MED) to determine total opioid medications given in the time period. MED is a standard conversion factor developed by the United States Centers for Disease Control and Prevention (CDC). The MED equates the many different opioids into a standard value that is based on morphine and its potency.
Time Frame: 0-4 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents (MME)
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 18
milligram morphine equivalents (MME) | 23.47 (20.74) | 37.89 (22.73)

14. Secondary Outcome: Opioid Consumption in Morphine Equivalent Dose 4-8 Hours Post-operative
Description: as for outcome 13
Time Frame: 4-8 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents (MME)
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 18
milligram morphine equivalents (MME) | 29.00 (26.91) | 39.94 (23.83)

15. Secondary Outcome: Opioid Consumption in Morphine Equivalent Dose 8-16 Hours Post-operative
Description: as for outcome 13
Time Frame: 8-16 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents (MME)
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 18
milligram morphine equivalents (MME) | 38.44 (34.04) | 52.53 (29.37)

16. Secondary Outcome: Opioid Consumption in Morphine Equivalent Dose 16-24 Hours Post-operative
Description: Post-operative opioid consumption in morphine equivalent dose (MED to determine total opioid medications given in the time period. MED is a standard conversion factor developed by the United States Centers for Disease Control and Prevention (CDC). The MED equates the many different opioids into a standard value that is based on morphine and its potency.
Time Frame: 16-24 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents (MME)
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 18
milligram morphine equivalents (MME) | 48.06 (44.36) | 64.64 (36.77)

17. Secondary Outcome: Opioid Consumption in Morphine Equivalent Dose 24-48 Hours Post-operative
Description: as for outcome 13
Time Frame: 24-48 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents (MME)
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 18
milligram morphine equivalents (MME) | 67.71 (65.83) | 92.64 (57.43)

18. Secondary Outcome: Opioid Consumption in Morphine Equivalent Dose 48-72 Hours Post-operative
Description: as for outcome 13
Time Frame: 48-72 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents (MME)
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 18
milligram morphine equivalents (MME) | 76.38 (80.33) | 105.61 (69.30)

19. Secondary Outcome: Total Intraoperative Opioid Consumption in Morphine Equivalent Dose
Description: Total opioids administered in morphine equivalent dose (MED) in the operating room during the surgery. MED is a standard conversion factor developed by the United States Centers for Disease Control and Prevention (CDC). The MED equates the many different opioids into a standard value that is based on morphine and its potency.
Time Frame: From start of surgery to end of surgery, an average of 2-3 hours
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents (MME)
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligram morphine equivalents (MME) | 63.1 (31.7) | 64.1 (35.4)

20. Secondary Outcome: Acetaminophen Consumption in Milligrams 0-4 Hours Post-operative
Description: Acetaminophen is a pain medication that is not an opioid. The acetaminophen use in milligrams will be compared in each group at different time points.
Time Frame: 0-4 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 679 (363) | 453 (459)

21. Secondary Outcome: Acetaminophen Consumption in Milligrams 4-8 Hours Post-operative
Description: as for outcome 20
Time Frame: 4-8 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 250 (358) | 329 (412)

22. Secondary Outcome: Acetaminophen Consumption in Milligrams 8-16 Hours Post-operative
Description: as for outcome 20
Time Frame: 8-16 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 988 (398) | 842 (462)

23. Secondary Outcome: Acetaminophen Consumption in Milligrams 16-24 Hours Post-operative
Description: as for outcome 20
Time Frame: 16-24 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 835 (513) | 900 (596)

24. Secondary Outcome: Acetaminophen Consumption in Milligrams 24-48 Hours Post-operative
Description: as for outcome 20
Time Frame: 24-48 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 2159 (1393) | 2676 (1699)

25. Secondary Outcome: Acetaminophen Consumption in Milligrams 48-72 Hours Post-operative
Description: as for outcome 20
Time Frame: 48-72 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 1385 (1391) | 1453 (1843)

26. Secondary Outcome: Gabapentin Consumption in Milligrams 0-4 Hours Post-operative
Description: Gabapentin is a pain medication that is not an opioid. The gabapentin use in milligrams will be compared in each group at different time points.
Time Frame: 0-4 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 58.82 (100.37) | 68.42 (149.27)

27. Secondary Outcome: Gabapentin Consumption in Milligrams 4-8 Hours Post-operative
Description: as for outcome 26
Time Frame: 4-8 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 52.94 (117.89) | 36.84 (76.09)

28. Secondary Outcome: Gabapentin Consumption in Milligrams 8-16 Hours Post-operative
Description: as for outcome 26
Time Frame: 8-16 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 82.35 (113.11) | 115.79 (167.54)

29. Secondary Outcome: Gabapentin Consumption in Milligrams 16-24 Hours Post-operative
Description: as for outcome 26
Time Frame: 16-24 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 100.00 (122.47) | 189.47 (196.91)

30. Secondary Outcome: Gabapentin Consumption in Milligrams 24-48 Hours Post-operative
Description: as for outcome 26
Time Frame: 24-48 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 223.53 (343.75) | 452.63 (505.93)

31. Secondary Outcome: Gabapentin Consumption in Milligrams 48-72 Hours Post-operative
Description: as for outcome 26
Time Frame: 48-72 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 152.94 (260.09) | 300.00 (458.26)

32. Secondary Outcome: Ketorolac Consumption in Milligrams 0-4 Hours Post-operative
Description: The ketorolac use in milligrams will be compared in each group at different time points.
Time Frame: 0-4 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 1.765 (7.276) | 2.895 (7.695)

33. Secondary Outcome: Ketorolac Consumption in Milligrams 4-8 Hours Post-operative
Description: The ketorolac use in milligrams will be compared in each group at different time points.
Time Frame: 4-8 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 3.529 (8.434) | 0.789 (3.441)

34. Secondary Outcome: Ketorolac Consumption in Milligrams 8-16 Hours Post-operative
Description: The ketorolac use in milligrams will be compared in each group at different time points.
Time Frame: 8-16 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 6.176 (10.684) | 5.789 (10.576)

35. Secondary Outcome: Ketorolac Consumption in Milligrams 16-24 Hours Post-operative
Description: The ketorolac use in milligrams will be compared in each group at different time points.
Time Frame: 16-24 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 0 (0) | 8.421 (11.432)

36. Secondary Outcome: Ketorolac Consumption in Milligrams 24-48 Hours Post-operative
Description: The ketorolac use in milligrams will be compared in each group at different time points.
Time Frame: 24-48 hours post-operative.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 17.647 (35.669) | 21.842 (26.416)

37. Secondary Outcome: Ketorolac Consumption in Milligrams 48-72 Hours Post-operative
Description: Ketorolac is a pain medication that is not an opioid. The ketorolac use in milligrams will be compared in each group at different time points.
Time Frame: 48-72 hours post-operative
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
milligrams | 11.471 (24.607) | 5.526 (14.327)

38. Secondary Outcome: Postoperative Quality of Recovery Score (QOR-15) 12-24 Hours Post-operative
Description: A survey on patient reported outcomes which consists of 15 questions related to five domains of patient reported health status (pain, physical comfort, physical independence, psychological support and emotional state). The score is reported on a scale from 0 to 150 with higher scores meaning a better outcome.
Time Frame: 12-24 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 12 | 9
score on a scale | 8.24 (0.96) | 7.29 (1.36)

39. Secondary Outcome: Postoperative Quality of Recovery Score (QOR-15) 24 to 48 Hours Post-operative
Description: as for outcome 38
Time Frame: 24-48 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 13 | 8
score on a scale | 8.26 (0.77) | 8.40 (0.86)

40. Secondary Outcome: Postoperative Quality of Recovery Score (QOR-15) 48 to 72 Hours Post-operative
Description: as for outcome 38
Time Frame: 48-72 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 6 | 4
score on a scale | 8.56 (0.90) | 8.52 (0.95)

41. Secondary Outcome: Post-operative Incentive Spirometry Changes From Preoperative Baseline at 0-4 Hours Post-operative
Description: Incentive spirometry measures how much air you can inhale, which can help indicate how well your lungs are working after surgery. Incentive spirometry measures the volume (or amount) of air you inhale measured in cubic centimeters (cc). Higher numbers indicate that you're inhaling more air. This measure will be the change in incentive spirometry from baseline (baseline incentive spirometry - incentive spirometry 0 to 4 hours post-operative). A negative number reflects reduced volume of air.
Time Frame: 0-4 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: volume of air in cubic centimeters
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 16 | 18
volume of air in cubic centimeters | -956.25 (528.796) | -652.778 (596.429)

42. Secondary Outcome: Post-operative Incentive Spirometry Changes From Preoperative Baseline at 4-8 Hours Post-operative
Description: Incentive spirometry measures how much air you can inhale, which can help indicate how well your lungs are working after surgery. Incentive spirometry measures the volume (or amount) of air you inhale measured in cubic centimeters (cc). Higher numbers indicate that you're inhaling more air. This measure will be the change in incentive spirometry from baseline (baseline incentive spirometry - incentive spirometry 4 to 8 hours post-operative). A negative number reflects reduced volume of air.
Time Frame: 4-8 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: volume of air in cubic centimeters
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 13 | 14
volume of air in cubic centimeters | -815.385 (632.582) | -775 (765.544)

43. Secondary Outcome: Post-operative Incentive Spirometry Changes From Preoperative Baseline at 8-12 Hours Post-operative
Description: Incentive spirometry measures how much air you can inhale, which can help indicate how well your lungs are working after surgery. Incentive spirometry measures the volume (or amount) of air you inhale measured in cubic centimeters (cc). Higher numbers indicate that you're inhaling more air. This measure will be the change in incentive spirometry from baseline (baseline incentive spirometry - incentive spirometry 8 to 12 hours post-operative). A negative number reflects reduced volume of air.
Time Frame: 8-12 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: volume of air in cubic centimeters
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 9 | 11
volume of air in cubic centimeters | -1005.556 (682.113) | -959.091 (654.912)

44. Secondary Outcome: Post-operative Incentive Spirometry Changes From Preoperative Baseline at 12-24 Hours Post-operative
Description: Incentive spirometry measures how much air you can inhale, which can help indicate how well your lungs are working after surgery. Incentive spirometry measures the volume (or amount) of air you inhale measured in cubic centimeters (cc). Higher numbers indicate that you're inhaling more air. This measure will be the change in incentive spirometry from baseline (baseline incentive spirometry - incentive spirometry 12 to 24 hours post-operative). A negative number reflects reduced volume of air.
Time Frame: 12-24 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: volume of air in cubic centimeters
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 15 | 15
volume of air in cubic centimeters | -718.333 (575.114) | -853.333 (747.01)

45. Secondary Outcome: Post-operative Incentive Spirometry Changes From Preoperative Baseline at 24-48 Hours Post-operative
Description: Incentive spirometry measures how much air you can inhale, which can help indicate how well your lungs are working after surgery. Incentive spirometry measures the volume (or amount) of air you inhale measured in cubic centimeters (cc). Higher numbers indicate that you're inhaling more air. This measure will be the change in incentive spirometry from baseline (baseline incentive spirometry - incentive spirometry 24 to 48 hours post-operative). A negative number reflects reduced volume of air.
Time Frame: 24-48 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: volume of air in cubic centimeters
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 14 | 17
volume of air in cubic centimeters | -975 (640.538) | -700 (537.936)

46. Secondary Outcome: Post-operative Incentive Spirometry Changes From Preoperative Baseline at 48-72 Hours Post-operative
Description: Incentive spirometry measures how much air you can inhale, which can help indicate how well your lungs are working after surgery. Incentive spirometry measures the volume (or amount) of air you inhale measured in cubic centimeters (cc). Higher numbers indicate that you're inhaling more air. This measure will be the change in incentive spirometry from baseline (baseline incentive spirometry - incentive spirometry 48 to 72 hours post-operative). A negative number reflects reduced volume of air.
Time Frame: 48-72 hours post-operative
Population: The number of participants analyzed differs across outcome measures due to incomplete data collection for some outcomes.
Measure: Mean (Standard Deviation); unit: volume of air in cubic centimeters
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 8 | 7
volume of air in cubic centimeters | -906.25 (651.612) | -642.857 (403.556)

47. Secondary Outcome: Length of Hospital Stay
Description: Number of hours from admission to discharge
Time Frame: From date of admission until date of discharge, an average of 72 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
Number analyzed (Participants) | 17 | 19
Hours | 72.00 [53.00 to 79.00] | 58.00 [55.00 to 77.50]

ADVERSE EVENTS:
Time Frame: From start of surgery to up to 72 hours post-operative
Description: Adverse events are reported for all randomized participants
Arm/Group | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine | Continuous Catheter Infusion Ropivacaine
All-Cause Mortality (participants affected / at risk) | 2/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/22
Other Adverse Events (participants affected / at risk) | 3/23 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine (N=23) | Continuous Catheter Infusion Ropivacaine (N=22)
Subcutaneous emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Intraoperative hemorrhage (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Shot Liposomal Bupivacaine (EXPAREL®)/Bupivacaine (N=23) | Continuous Catheter Infusion Ropivacaine (N=22)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Pain of skin (Surgical and medical procedures) | 1 | 1 (1) — Pain at injection site
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04559347/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT04559347/SAP_001.pdf